CLINICAL TRIAL: NCT01436422
Title: A Phase 1 Evaluation of the Safety and Immunogenicity of the Recombinant Live Attenuated Tetravalent Dengue Virus Vaccine Admixtures TV003 and TV005 in Healthy Flavivirus-Naïve Adult Subjects
Brief Title: Evaluating the Safety and Immune Response to Two Admixtures of a Tetravalent Dengue Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 279
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Dengue
Keywords: Dengue Virus; Dengue Fever; Dengue Vaccine; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TetraVax-DV Vaccine - Admixture TV003 (Experimental): Participants will receive the TetraVax-DV Vaccine - Admixture TV003 at Day 0 and Day 180.
  Interventions: Biological: TetraVax-DV Vaccine - Admixture TV003
- TetraVax-DV Vaccine - Admixture TV005 (Experimental): Participants will receive the TetraVax-DV Vaccine - Admixture TV005 at Day 0 and Day 180.
  Interventions: Biological: TetraVax-DV Vaccine - Admixture TV005
- Placebo (Placebo Comparator): Participants will receive the placebo at Day 0 and Day 180.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV Vaccine - Admixture TV003 — One subcutaneous injection at Day 0 and Day 180 of a live attenuated recombinant TetraVax-DV vaccine, Admixture TV003 (10^3 PFU of rDEN1Δ30, 10^3 PFU of rDEN2/4Δ30(ME), 10^3 PFU of rDEN3Δ30/31-7164, and 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine - Admixture TV003
Biological: TetraVax-DV Vaccine - Admixture TV005 — One subcutaneous injection at Day 0 and Day 180 of a live attenuated recombinant TetraVax-DV vaccine, Admixture TV005 (10^3 PFU of rDEN1Δ30, 10^4 PFU of rDEN2/4Δ30(ME), 10^3 PFU of rDEN3Δ30/31-7164, and 10^3 PFU of rDEN4Δ30)
  Arms: TetraVax-DV Vaccine - Admixture TV005
Biological: Placebo — One subcutaneous injection at Day 0 and Day 180 of placebo
  Arms: Placebo

SUMMARY:
Dengue viruses can cause dengue fever and other serious health conditions, primarily affecting people living in tropical regions of the world. This study will evaluate the safety and immune responses to two formulations of a tetravalent dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever and the more severe condition, dengue hemorrhagic fever/shock syndrome. Dengue viruses are common in most tropical and subtropical regions of the world and infection with dengue viruses is the leading cause of hospitalization and death in children in many tropical Asian countries. For these reasons, the World Health Organization (WHO) has made the development of a dengue virus vaccine a top priority. This study will evaluate the safety and immunogenicity of two doses of a live, attenuated, tetravalent dengue virus vaccine called TetraVax-DV in healthy adults. Two different versions of the TetraVax-DV vaccine will be evaluated.

This study will enroll healthy adults 18-50 years old. Participants will be randomly assigned to receive one of two admixtures of the TetraVax-DV vaccine or a placebo. At a baseline study visit, participants will undergo a medical history review, physical examination, blood collection, vital sign measurements, and a pregnancy test for females. Participants will then receive one injection of their assigned vaccine in the upper arm. After receiving the vaccine, participants will remain in the clinic for 30 minutes for observation and monitoring. At home, participants will monitor and record their temperature three times a day for 16 days. Additional study visits will occur at Days 3, 8, 10, 12, 14, 16, 21, 28, 56, 90, and 150 and will include a physical examination, assessment of symptoms, and blood collection. On Day 180, participants will receive a second injection of the same vaccine they received at the baseline study visit. Follow-up study visits will occur at Days 183, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360, and will include the same study procedures and monitoring that occurred after the first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-vaccination
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Currently pregnant (as determined by positive beta-human choriogonadotropin [HCG] test) or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in the protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the 12 months prior to study entry that has caused medical, occupational, or family problems, as indicated by a participant's history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the 6 months prior to study entry)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Asplenia
* Receipt of blood products within the 6 months prior to study entry, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Inclusion Criteria for Second Dose of Vaccine:

* In good general health, as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 6 months post-vaccination
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must be willing to use effective contraception for the duration of the trial. More information on this criterion can be found in the protocol.

Exclusion Criteria for Second Dose of Vaccine:

* Anaphylaxis or angioedema following the first dose of vaccine
* Currently pregnant (as determined by positive beta-HCG test) or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the 12 months prior to study entry which has caused medical, occupational, or family problems, as indicated by a participant's history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the 6 months prior to study entry)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV) infection, by hepatitis B surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 42 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 42 days following vaccination
* Asplenia
* Receipt of blood products within the 6 months prior to study entry, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 42 days following vaccination
* Anticipated receipt of any other investigational agent in the 42 days before or after vaccination
* Has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Other Treatments and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

Ongoing Exclusion Criteria:

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 42-day period post-vaccination
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 42-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 42-day period post-vaccination
* Receipt of immunoglobulins and/or any blood products during the 42-day period post-vaccination
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety of two TetraVax-DV admixtures, as assessed by the frequency of vaccine-related adverse events (AEs), graded by severity | Measured through Day 360
Immunogenicity of two TetraVax-DV admixtures, as assessed by neutralizing antibody titers to DEN1, DEN2, DEN3, and DEN4 | Measured through Day 180 after each vaccination
  Monovalent, bivalent, trivalent, and tetravalent seropositivity and seroconversion rates will be determined at 28, 56, and 90 days after each vaccination.
Seropositivity in those vaccinees who remained seronegative to one or more DENV serotypes following the first vaccination and who recieved a second dose of vaccine given at Day 180 | Measured through Day 360

SECONDARY OUTCOMES:
Frequency of viremia following vaccination | Measured through Day 360
Number of vaccinees infected with DEN1, DEN2, DEN3, and DEN4 | Measured through Day 360
  Infection is defined as recovery of vaccine virus from the blood or serum of a participant and/or by seropositivity to DEN virus (PRNT50 greater than or equal to 1:10).
Duration of the neutralizing antibody response 26 weeks after each vaccination | Measured 26 weeks after each vaccination
Ability of a second dose of vaccine to boost serum neutralizing antibody titers by Day 270 | Measured at Day 270
  Boost will be defined as a greater than or equal to 4-fold rise in serum neutralizing antibody titer by Day 270 compared with Day 180.
Evaluate the phenotype of peripheral blood mononuclear cells at primary infection with the TetraVax-DV vaccine | Measured through Day 360
Evaluate the cellular immune response to primary infection with the TetraVax-DV vaccine | Measured through Day 360
Evaluate the innate immune response to primary infection with the TetraVax-DV vaccine | Measured through Day 360
Evaluate B and T cell memory responses following primary and secondary infections with TetraVax-DV vaccine | Measured through Day 360
Quantity of viremia following vaccination | Measured through Day 360
Duration of viremia following vaccination | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (3):
- United States (3):
  - Center for Immunization Research, Johns Hopkins School of Public Health, Baltimore, Maryland
  - Fletcher Allen Health Care (FAHC), General Clinical Research Center (GCRC), Burlington, Vermont
  - University of Vermont Vaccine Testing Center, Burlington, Vermont

REFERENCES:
- [Background] Bhamarapravati N, Sutee Y. Live attenuated tetravalent dengue vaccine. Vaccine. 2000 May 26;18 Suppl 2:44-7. doi: 10.1016/s0264-410x(00)00040-2. PMID 10821973
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Durbin AP, Kirkpatrick BD, Pierce KK, Schmidt AC, Whitehead SS. Development and clinical evaluation of multiple investigational monovalent DENV vaccines to identify components for inclusion in a live attenuated tetravalent DENV vaccine. Vaccine. 2011 Sep 23;29(42):7242-50. doi: 10.1016/j.vaccine.2011.07.023. Epub 2011 Jul 21. PMID 21781997
- [Derived] Kirkpatrick BD, Durbin AP, Pierce KK, Carmolli MP, Tibery CM, Grier PL, Hynes N, Diehl SA, Elwood D, Jarvis AP, Sabundayo BP, Lyon CE, Larsson CJ, Jo M, Lovchik JM, Luke CJ, Walsh MC, Fraser EA, Subbarao K, Whitehead SS. Robust and Balanced Immune Responses to All 4 Dengue Virus Serotypes Following Administration of a Single Dose of a Live Attenuated Tetravalent Dengue Vaccine to Healthy, Flavivirus-Naive Adults. J Infect Dis. 2015 Sep 1;212(5):702-10. doi: 10.1093/infdis/jiv082. Epub 2015 Mar 22. PMID 25801652